CLINICAL TRIAL: NCT04437030
Title: Multiparametric Photoacoustic Imaging in the Course of Radiation Therapy of Malignant Head and Neck Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Juergen Debus, Head of Department, University Hospital Heidelberg
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MSOT HNC
Record Dates: First submitted 2020-06-09; First posted 2020-06-18 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient (Active Comparator): Patient with Head and neck cancer
  Interventions: Device: MSOT Acuity Echo device
- Healthy subjects (Other): Healty subjects with not history of Tumor disease in the Head and neck region
  Interventions: Device: MSOT Acuity Echo device

INTERVENTIONS:
Device: MSOT Acuity Echo device — The MSOT acutiy Echo device can take ultrasound recordings in addition to photoacoustic recordings.

SUMMARY:
Multispectral photoacoustic imaging enables the measurement of the optical absorption of various tissue components or exogenous contrast agents in vivo. The dominant, near infrared absorbing chromophores in human tissue are oxy- and deoxyhemoglobin followed by collagen, melanin and lipids. The multispectral measurement of the absorption of hemoglobin shows changes in blood oxygen saturation and blood volume. The high resolution of photoacoustic imaging also enables the vascular structure to be displayed. The aim of this exploratory study is to generate hypotheses by applying photoacoustic imaging to the field of head and neck tumor therapy. The next step is to investigate whether and how photoacoustic imaging can help improve diagnostics and better planning of treatments in the future. In particular, the differences between normal and tumor tissue and the changes in the tissue due to radiation therapy using photoacoustic imaging are examined. In the quantitative analysis of the images, measured chromophores, primarily oxygen saturation, blood volume and collagen concentrations at different measuring points are used in the course of the therapy.

DETAILED DESCRIPTION:
Multispectral photoacoustics enable non-invasive, inexpensive and dose-free real-time imaging of light-absorbing molecules (absorbers), e.g. Deoxyhemoglobin and oxygenated hemoglobin in human tissue. This allows blood oxygen saturation (sO2) to be determined at depths of up to several centimeters. Measurements of correlates to blood volume and collagen concentration are also made possible. In photoacoustic imaging, the tissue to be examined is irradiated with nanosecond short, near-infrared (650 - 1300nm) laser pulses. If laser light is locally absorbed by a tissue structure, it expands thermoelastically, which triggers an ultrasonic pressure wave, which is measured with the aid of an ultrasonic head. The initial pressure distribution and thus the absorption in the tissue can then be reconstructed. Since different molecules show distinct absorption behavior depending on the wavelength in the near infrared, by acquiring several wavelengths it is possible to estimate which absorbers are in which concentration in a tissue structure. The effectiveness and tolerability of modern high-precision radiation therapy for head and neck tumors largely depends on the quality of the imaging. The potential diagnostic benefits of photoacoustics in the radiotherapy of patients with head and neck tumors principally concern the target volume definition, the implementation of image-guided, adaptive radiotherapy and imaging tumor follow-up as well as the early detection of tumors.

Multispectral photoacoustics primarily enable the analysis of tumor hypoxia, which has been associated several times with increased radio resistance and an unfavorable prognosis. In addition, other factors, e.g. the blood volume and the collagen content in the tissue are analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness and ability to participate
2. sufficient knowledge of German to understand the patient / subject information and the declaration of consent,
3. tumor disease to be treated by radiotherapy in the neck and neck area,
4. Completed wound healing after operative interventions in the head and neck area,
5. The patient's consent and written consent,
6. the patient's ability to assess the nature and scope as well as possible consequences of the clinical study,

8. Age ≥ 18 years.

Requirement 3 does not apply to the control group of healthy subjects

Exclusion Criteria:

* Pre-radiation in the head and neck area
* Inadequate regression of toxicities from previous therapies
* Indications that the participant is unlikely to adhere to the study protocol (e.g. lack of compliance)
* Missing written declaration of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
diagnostic feasibility of photoacoustic imaging: Oxygen Saturation | previouse to Radiotherapy start
  Measurement of Oxygen Saturation in the tumor tissue
diagnostic feasibility of photoacoustic imaging: Oxygen Saturation | 3 weeks after Radiotherapy start
  Measurement of Oxygen Saturation in the tumor tissue
diagnostic feasibility of photoacoustic imaging: Oxygen Saturation | 3 month after Radiotherapy start
  Measurement of Oxygen Saturation in the tumor tissue
diagnostic feasibility of photoacoustic imaging: blood volume | previouse to Radiotherapy start
  blood volume
diagnostic feasibility of photoacoustic imaging: blood volume | 3 weeks after Radiotherapy start
  blood volume
diagnostic feasibility of photoacoustic imaging: blood volume | 3 month after Radiotherapy start
  blood volume
diagnostic feasibility of photoacoustic imaging: blood volume | previouse to Radiotherapy start
  amount of collagen in the tumor tissue
diagnostic feasibility of photoacoustic imaging: amount of collagen in the tumor tissue | 3 weeks after Radiotherapy start
  amount of collagen in the tumor tissue
diagnostic feasibility of photoacoustic imaging: amount of collagen in the tumor tissue | 3 month after Radiotherapy start
  amount of collagen in the tumor tissue

SECONDARY OUTCOMES:
Analysis of Tumor tissue and normal tissue | previouse to Radiotherapy start
  Differences of Oxygen saturation
Analysis of Tumor tissue and normal tissue | 3 weeks after Radiotherapy start
  Differences of Oxygen saturation
Analysis of Tumor tissue and normal tissue | 3 month after Radiotherapy start
  Differences of Oxygen saturation
Analysis of Tumor tissue and normal tissue | previouse to Radiotherapy start
  blood volume
Analysis of Tumor tissue and normal tissue | 3 weeks after Radiotherapy start
  blood volume
Analysis of Tumor tissue and normal tissue | 3 month after Radiotherapy start
  blood volume
Analysis of Tumor tissue and normal tissue | previouse to Radiotherapy start
  amount of collagen
Analysis of Tumor tissue and normal tissue | 3 weeks after Radiotherapy start
  amount of collagen
Analysis of Tumor tissue and normal tissue | 3 month after Radiotherapy start
  amount of collagen
multimodal information about tissue morphology | previouse to Radiotherapy start
  Registration of photoaccustic and MRI/CT Imaging
multimodal information about tissue function | 3 weeks after Radiotherapy start
  Registration of photoaccustic and MRI/CT Imaging
multimodal information about tissue function | 3 month after Radiotherapy start
  Registration of photoaccustic and MRI/CT Imaging

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Adeberg, PD, Principal Investigator — University Hospital Heidelberg
Locations (1):
- University Hopsital Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No